CLINICAL TRIAL: NCT01672580
Title: Diffusion of Health Interventions Across Social Networks in Honduran Villages
Brief Title: Social Network Interventions in Rural Honduras
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Thomas Keegan, Ph.D., Project Director, Yale University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Lempira_Phase2
Record Dates: First submitted 2012-08-20; First posted 2012-08-27 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Malnutrition; Dysentery; Social Transmission of Health Behaviors
Keywords: social networks; nutrition; vitamins; chlorine
MeSH Terms: conditions — Malnutrition; Dysentery | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Random-Cloro (Active Comparator): exposure to water chlorination
  Interventions: Behavioral: exposure to water chlorination
- Random-Vitamin (Active Comparator): exposure to vitamin use
  Interventions: Behavioral: exposure to vitamin use
- Indegree-Cloro (Experimental): high in-degree, exposure to water chlorination
  Interventions: Behavioral: exposure to water chlorination; Behavioral: high in-degree
- Indegree-Vitamin (Experimental): high in-degree, exposure to vitamin use
  Interventions: Behavioral: exposure to vitamin use; Behavioral: high in-degree
- Nominated-Cloro (Experimental): nominated by random, exposure to water chlorination
  Interventions: Behavioral: exposure to water chlorination; Behavioral: nominated by random
- Nominated-Vitamin (Experimental): nominated by random, exposure to vitamin use
  Interventions: Behavioral: exposure to vitamin use; Behavioral: nominated by random

INTERVENTIONS:
Behavioral: exposure to vitamin use — "Seed" individuals in village are given daily adult multivitamin, with training on use and general nutrition information, along with coupons to distribute to others in village
  Other Names: Medox Forte
  Arms: Indegree-Vitamin; Nominated-Vitamin; Random-Vitamin
Behavioral: exposure to water chlorination — "Seed" individuals in village are given Clorox bleach for water purification, with training on use and general information on water hygiene, along with coupons to distribute to others in village
  Other Names: Clorox
  Arms: Indegree-Cloro; Nominated-Cloro; Random-Cloro
Behavioral: high in-degree — "Seed" individuals for starting intervention are chosen on the basis of high (social network) in-degree
  Arms: Indegree-Cloro; Indegree-Vitamin
Behavioral: nominated by random — "Seed" individuals for starting intervention are chosen on the basis of being named as a friend/alter of a randomly selected individual
  Arms: Nominated-Cloro; Nominated-Vitamin

SUMMARY:
This project will examine the spread of health interventions with a randomized control trial design by introducing public health interventions in 32 villages in the Honduran Department of Lempira. Based on identified public health needs in the region, namely improved drinking water and diet, this study will provide training on the use of chlorine (sodium hypochlorite) for water purification and multivitamins for nutritional supplementation. In some villages, individuals selected for their social connectedness will be trained and given coupons that can be redeemed for either chlorine bleach or multivitamins, and these persons will be asked to spread this information and distribute coupons to four people of their choosing. In other villages, individuals selected at random will receive the same training, materials, and instructions. A second wave of coupon distribution will provide coupons to those who received a coupon from the original "seed" groups so that they may disperse these coupons further out in the social networks. Over the following months, study investigators will look at how knowledge of these health practices, and uptake or and adherence to the practices, spreads throughout the villages.

More specifically, the investigators will examine the speed and extent of spreading of these new health practices after introducing them to three different initial "seed" groups: (1) people chosen on the basis of being named as a friend by many people in their village, (2) people chosen based on being named as a friend by a randomly chosen individual, and (3) a group of randomly chosen individuals. It is hypothesized that spread will occur faster and/or to a greater extent when the intervention is started in groups 1 and 2 versus group 3 (control group).

ELIGIBILITY:
Inclusion Criteria:

* Residents of Targeted Communities, ages 15 and up

Exclusion Criteria:

* Children younger than age 15

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5773 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Intervention Spread | October 2012
  Use of health product among community members will be tracked.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Christakis, MD, PhD, Principal Investigator — Yale University; Thomas Keegan, PhD, Study Director — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Kim DA, Hwong AR, Stafford D, Hughes DA, O'Malley AJ, Fowler JH, Christakis NA. Social network targeting to maximise population behaviour change: a cluster randomised controlled trial. Lancet. 2015 Jul 11;386(9989):145-53. doi: 10.1016/S0140-6736(15)60095-2. Epub 2015 May 4. PMID 25952354